CLINICAL TRIAL: NCT00146718
Title: Anti-malarial Drug Resistance in Cameroon: Therapeutic Efficacy and Biological Markers of Resistance
Brief Title: Anti-Malarial Drug Resistance in Cameroon
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: University of Yaounde (Other)
Responsible Party: Principal Investigator, Brian Greenwood, Professor, London School of Hygiene and Tropical Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ITDCVG34
Record Dates: First submitted 2005-09-05; First posted 2005-09-07 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2017-01

CONDITIONS: Malaria
Keywords: malaria; drug resistance; antimalarials
MeSH Terms: conditions — Malaria | interventions — Amodiaquine; Sulfadoxine; Pyrimethamine

INTERVENTIONS:
Drug: Amodiaquine and Sulphadoxine/Pyrimethamine

SUMMARY:
The project is a three-armed study designed to evaluate the efficacy of amodiaquine(AQ), sulphadoxine-pyrimethamine(SP) and(AQ+SP) in three sites in Cameroon that differ in their baseline characteristics for malaria. In addition, drug resistance will be determined by measurement of blood drug levels,and identification of molecular markers of resistance.

DETAILED DESCRIPTION:
The objectives of this study are:- .

* to evaluate the therapeutic efficacy of amodiaquine(AQ), Fansidar(SP) and the combination amodiaquine/Fansidar in three sites in Cameroon namely, Garoua (Sahel-savanna), Yaounde (Forest-savannah mosaic) and Limbe (Littoral-forest)
* to determine the prevalence of molecular markers associated with resistance to chloroquine,AQ,and SP in Limbe and Garoua and of mefloquine in Yaounde.
* to investigate biological factors that may enhance anti-malaria therapeutic efficacy. This will involve an exploratory, pilot study conducted during the second year of the program.

Patients will be rapidly screened for temperature and sent to the laboratory to determine the presence or absence of malaria parasites. The patients will then be examined clinically for inclusion or exclusion. Consent will be sort from the parents and the children randomised and assigned study numbers. To avoid bias in assigning the patients to groups and to ensure equal numbers in the treatment groups, blocked randomization will be performed, using a table of random variables of varying block sizes. The physician is blinded to what treatment the patient gets.

Amodiaquine will be administered at 10mg/kg on each of the three days to children in the AQ treatment group, together with Fansidar dummy tablets. Fansidar will be given at 25 mg/kg on day 0 and quinine as rescue drug at 10mg/kg per 8H for 6 days. For the AQ/SP combination, on D0, patients will be given both 25 mg/kg SP and 10mg/kg AQ. On subsequent days the AQ or its dummy tablets(SP arm) will be given.

Clinical assessment during the study will include: physical examination and monitoring of vital signs on D0, D3, D7, D14 and D28. Hematological measurements will include: blood films, haemoglobin,glucose,blood drug levels,and baseline haematology. A maximum of 3ml of blood will be withdrawn from the patients in Yaoundé for complete analyses(see below). For patients recruited at Limbe and Garoua only finger prick blood filter paper samples will be obtained.

Day 0 blood samples (3mL) will be collected aseptically by venepuncture before therapy from each of 50 patients in Yaoundé using acid-citrate-dextrose buffer (ACD) as anticoagulant. This will be processed to provide plasma for immunological determinations and for haematology and blood drug level determinations.

The molecular characterization of diversity and mutations:

* the genetic heterogeneity of the study population will be established using primers for msp1 and msp2 shown previously to distinguish between strains.
* PCR products will be digested with restriction enzyme (RFLP-PCR) for pyrimethamine resistance genes dhfr and dhps, and for chloroquine resistant strains of the pfcrtgene.

ELIGIBILITY:
Inclusion criteria:

* Children 6-59 months of age
* Recorded temperature between 37.5oC and 39.5 oC
* Signs/symptoms of acute uncomplicated P. falciparum malaria.
* Positive microscopy for mono-infection with P falciparum malaria
* Asexual blood stage parasitaemia in the range 1,000 to 100,000 asexual parasites per ul
* Consent from parent or guardian of a child.
* No other apparent cause for the child's illness.

Exclusion criteria:

* Presence of signs of severe complicated falciparum malaria.
* Cerebral malaria (unrousable coma)
* Vomiting > twice within preceding 24 hours
* More than one convulsion within preceding 24 hours
* Inability to drink or breast-feed, or to take oral medication
* Haemoglobin less than 5g/dl or a hematocrit of less than 15%.
* Documented evidence of adequate treatment with drugs expected to be effective in the preceding 72 hours
* Presence of underlying diseases (cardiac, renal, hepatic,malnutrition, gastrointestinal)
* History of allergy to study drug
* Inability to attend for the stipulated follow-up visits,
* Difficulty in accessing the health facility, or any situation or condition which may compromise the patients ability to comply with the trial procedures.

Ages: 6 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 755
Dates: Start 2003-08; Study Completion 2005-05

PRIMARY OUTCOMES:
Adequate clinical and parasitological response(ACPR) on Day 28

SECONDARY OUTCOMES:
ACPR Day 14
Early treatment failure, between days 1 and 3
Late treatment failure, between days 4 and 14

CONTACTS AND LOCATIONS:
Overall Officials: Wilfred Mbacham, ScD, Principal Investigator — Laboratory for Public Health Biotechnology, University of Yaounde I